CLINICAL TRIAL: NCT04263116
Title: Balloon-Assisted Maturation of Autogenous Arteriovenous Fistulae; Clinical Efficacy and Complications: Randomized Prospective Study
Brief Title: Balloon-Assisted Maturation of Autogenous Arteriovenous Fistulae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R. 17.12.44
Record Dates: First submitted 2020-02-04; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Hemodialysis Access Failure

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Block randomization
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAM group (Experimental): Balloon assisted maturation
  Interventions: Procedure: Balloon Assisted Maturation
- NO BAM (Experimental): NO Balloon assisted maturation
  Interventions: Procedure: Balloon Assisted Maturation

INTERVENTIONS:
Procedure: Balloon Assisted Maturation — Angioplasty was performed under direct vision with or without the use of a guidewire using a 1 mm larger balloon than the size of the vein. BAM is performed over the whole length of the vein sparing the spatulated end of the vein

SUMMARY:
Background: There are several studies that document the safety and efficacy of the balloon-assisted maturation (BAM) technique. Ultimately, there are also studies that report its possible negative consequences such as fibrosis and restenosis of venous outflow, leading to malfunctioning arteriovenous fistula (AVF). Thus, in an effort to increase the number of primary AVFs, shorten maturation times, and reduce the number of indwelling catheters, we ascertain the BAM technique within this study to optimize access care and maximize use of AVFs. The balloon assisted maturation approach specifically and aggressively dilates the entire usable segment of the AVF.

Methods: This is a randomized prospective study conducted in the department of vascular surgery, Mansoura University Hospitals, including patients with hemodialysis access creation between June 2017 and May 2019. Three hundred patients were recruited from a total of 648 primary AVF creation cases. Patients were divided into two groups; Group (A) Balloon assisted maturation (BAM) (n=157) 52.3 % technique had been done while in the other Group (B) the usual maneuver was used (NO BAM) (n=143) 47.7%. Preoperative duplex was done for all cases to assess suitability. Intraoperative venography was the initial step following surgical exposure of the assigned veins to ascertain continuity and unlimited flow of the superficial vein. Balloon dilatation by 1 mm larger than the size of the vein, sparing the spatulated end of the vein followed by post-dilatation venography to reveal any injury and assess the success of dilatation process. All cases were completed as an end to side anastomosis. Patients were followed clinically and radiologically at regular visits in the 2nd, 4th and 6th week post-procedure, assessing the flow rate, vein depth and diameter via duplex US examination.

Results: Patients age ranged from 19 to 89 (mean 51.17 ±15.5) years. The average maturation time was 3.7 weeks (SD ± 1.3 w) and 5.91 weeks (SD ± 2.2 w) for the BAM and non-BAM groups, respectively. Eighty-seven cases (88.7 %) with a pre-operative vein diameter of 3 mm or less, that underwent BAM showed early maturation and started dialysis within 2-4 weeks (68 cases 70%). On the other hand, 28 cases (45.2%) with a vein diameter equal or less than 3 mm in the NO BAM group failed to get mature. Both successful functional maturation (95%) and complication rates (9.6 %) were higher among cases of the BAM group compared to 80.4% maturation rate and 5 % complication in the NO BAM group. The higher complication rate may be attributed to the large number of cases.

Conclusion: Balloon-assisted maturation has a pivotal role to help the dialysis society meet the goals of the Fistula First Initiative; It can achieve an accelerated functional maturation of AVF in cases of small caliber veins, with access to early dialysis, thus decreasing the indwelling catheter-related complications.

DETAILED DESCRIPTION:
INTRODUCTION:

End-stage renal disease (ESRD) is the crossing point of multiple heterogeneous disease pathways that can alter the structure and function of the kidneys irreversibly. Both definition and classification of ESRD have been developing over time. However, current international guidelines define ESRD as declined kidney function shown by GFR of less than 60 mL/min per 1•73 m², kidney damage markers or both, for at least 3 months duration, regardless of underlying cause.1 Haemodialysis (HD) is a lifeline management for patients with ESRD. A critical factor in the survival of renal dialysis patients is the surgical creation of vascular access, and international guidelines recommend arteriovenous fistulas (AVF) as the gold standard vascular access for haemodialysis. Arteriovenous graft and central vein catheters have higher primary patency rates compared to AVF, however native AVFs last longer. 3 There is conflicting evidence about the impact of various demographic characteristics of the patients on the functional maturation of the native AVFs. Certain characteristics such as diabetes mellitus, female gender, thrombophilia and various hematological factors, such as platelet count and hemoglobin levels, can affect fistula maturation. Also the impact of certain operative and anatomical factors, including but not limited to diameter of artery and venous limb of the AVF, presence of palpable thrill, audible bruit, and anatomical site of fistula may affect outcome.4 Functional fistula maturation is defined as patent fistula, ready for cannulation with vein length of at least 10 cm long segment, diameter more than 6 mm, depth not more than 6 mm and ability of the access to deliver a flow rate of 350 to 400 ml/min and maintain dialysis for 3.5 to 4 hours.5 Delayed maturation of AVF among patients who require hemodialysis can lead to catheter sepsis with its resultant morbidity and mortality. Some authors have proposed that sequential BAM may accelerate maturation process and shorten the maturation times of these accesses.6 Balloon angioplasty maturation is emerging as a surgical technique that could increase utilization and improve function of autogenous arteriovenous hemodialysis accesses. This approach includes primary balloon angioplasty (PBA) of small veins during AVF creation.9-10 However there are no studies that directly compare maturation times for AVF with and without using BAM. There are several studies that document the safety and efficacy of the BAM technique. 7 Ultimately, there are also studies that report its possible negative consequences such as fibrosis and restenosis of venous outflow, leading to malfunctioning AVF. 8 Thus, in an effort to increase the number of primary AVFs, shorten maturation times, and reduce the number of indwelling catheters, we ascertain the BAM technique within this study to optimize access care and maximize use of AVFs.

Patients and Methods:

This is a randomized prospective study conducted in the department of vascular surgery, Mansoura university hospitals. Between July 2017 and May 2019 Three hundred patients were recruited from a total of 648 primary AVF creation cases. Patients had been advised to undergo elective surgery for AVF once their renal glomerular filtration rate estimated (eGFR) is less than 15 ml/min. Block randomization was the method used for stratification of patients' groups.

Inclusion and exclusion criteria: All patients aged 18 years or older who need AVF formation in the upper limb were included as a recruitment target. In patients with multiple episodes of AVF creation, each episode was considered separately and data from the corresponding episode had been recorded in our data sheet. Patients who underwent salvage procedures to improve maturation, i.e. secondary maturation, or those who could not give informed consent were not included1. A total of 335 patients who needed Autogenous AVF were enrolled in the study during that period.

Patients and methods Table (1) shows the patient's demographics, including underlying medical conditions, previous AVF, transplanted kidney and other associated morbidity. Arterial assessments included pulse examination, segmental blood pressures in both upper extremities, and the modified Allen test for continuity of the palmar arch. Venous assessments include gross evaluation of the veins in the dependent position with tourniquet enhancement in the upper arm. Table (2) shows patients' workup including blood picture, blood sugar level, kidney functions, liver functions and coagulation profile.

Duplex US examination checked the diameter, compressibility, depth, and continuity of the arm veins. Arterial assessment included radial and brachial arterial size, presence or absence of calcification, segmental pressure, and velocity wave forms.

Operative procedure:

The non dominant upper limb was preferred and saved. AVFs were created at wrist, forearm and arm in both male and female patients under local, regional or general anaesthesia. All brachiobasilic fistulas were created in one stage.

Randomization was done through computer generated block serials in sealed envelopes which were opened when the patient was on the operating table. During AVF creation and before anastomosis, the vein was cannulated through the open end of the venotomy. Intraoperative venography was done to assess the vein in the BAM group only. Angioplasty was performed under direct vision with or without the use of a guidewire using a 1 mm larger balloon than the size of the vein. BAM is performed over the whole length of the vein sparing the spatulated end of the vein. Post venoplasty venography was done to reveal any injury and assess the dilatation process. All cases were completed as an end to side anastomosis followed by assessment of the dilated segment for any spasm which is treated by mechanical compression of the vein cephalad to the area of concern. Patients were discharged home on the following day with instructions for care of fistula.These instructions included avoidance of any blood sampling, using this arm for blood pressure measurement, clothes with constrictive sleeves, heavy or tight jewellery, circumferential dressings on wound and sleeping on the operated arm. Patients were taught how to feel for the thrill, advised to contact the operating team if they developed any numbness in hand, discoloration of fingertips or coldness. All patients were instructed to commence active hand ball exercises before discharge from hospital. Patients were followed both clinically and radiologically with duplex scan at the 2nd, 4th and 6th weeks post-procedure, checking the flow rate, depth and diameter of the target vein.

Statistical analysis: Data was analysed using Statistical Package for the Social Sciences. The numerical outcomes e.g. age was calculated as mean. Chi Square test was used to assess the association of various parameters. Results were considered statistically significant if the p-value was found to be less than or equal to 0.05. Log rank test (mantel cox) test was used to compare AVF maturation in both groups

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Any patient who need arterio-venous fistula formation in the upper limb

Exclusion Criteria:

* Patients who underwent salvage procedures to improve maturation, i.e. secondary maturation
* Those who could not give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2019-05-25 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Flow rate of the target vein | 6 weeks
  Radio-logically measure the flow rate in the vein
Diameter of the target vein | 6 weeks
  Radio-logically measure the vein diameter
Depth of the target vein | 6 weeks
  Radio-logically measure the vein depth from the skin

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No